CLINICAL TRIAL: NCT04890756
Title: Validity and Reliability of the Greek Version of the Modified Baecke Questionnaire
Brief Title: The Greek Version of Modified Baecke Questionnaire
Status: Completed | Type: Observational
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Vasiliki Stefanouli, Clinical Researcher, University of Thessaly
Other Study IDs: cepr_lab
Record Dates: First submitted 2021-04-22; First posted 2021-05-18 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Physical Activity
Keywords: validation; reliability; adaptation; questionnaire; Greek version; Baecke
MeSH Terms: conditions — Motor Activity | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Reliability Group: 100 Healthy Adults
  Interventions: Other: observational
- Validity Group: 45 Healthy Adults
  Interventions: Other: observational

INTERVENTIONS:
Other: observational — The reliability was determined (n=100) by filling out the mBQ, two times, one week apart (test-retest).
  For validation (n=45), the scores between the modified Baecke Questionnaire and the International Physical Activity Questionnaire were compared and the correlation between the modified Baecke Questionnaire and VO2max(via Astrand-Rhyming Cycle Ergometer Test) and between mBQ and interview (via METS) were assessed.

SUMMARY:
The purpose of this study was to translate and investigate the validity and reliability of the modified Baecke Physical Activity Questionnaire (mBQ) in the Greek adult population.

DETAILED DESCRIPTION:
The purpose of this study was to translate and investigate the validity and reliability of the modified Baecke Physical Activity Questionnaire (mBQ) in the Greek adult population. The cross-cultural adaptation of the mBQ was performed according to official guidelines.The reliability was determined by filling out the mBQ, two times, one week apart. For validation, the scores between the mBQ and the IPAQ were compared and the correlation between mBQ and VO2max and between mBQ and interview (METS) were assessed.

ELIGIBILITY:
Inclusion Criteria:

1. age above 18
2. Greek native speakers
3. Greek inhabitants
4. sufficient cognitive functioning.

Exclusion Criteria:

1. poor health status,
2. diagnosed with cardiovascular diseases
3. cardiac pacemaker,
4. medication that prevents exercise activity
5. neurological disorders with effect on the lower body
6. musculoskeletal disorders or injuries on the lower body in the last 3 months
7. PAR-Q health risk assessment form

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy
Sampling Method: Probability Sample
Enrollment: 145 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2016-07-20 (Actual); Study Completion 2021-03-25 (Actual)

PRIMARY OUTCOMES:
Reliability | one week apart
  The reliability was determined by filling out the modified Baecke Questionnaire, two times, one week apart (test-Retest).
  Tool: Modified Baecke Questionnaire (test-retest)
Validity | 1) IPAQ ( Time Frame: 30 min) 2) Astrand-Rhyming Cycle Ergometer Test (Time Frame: 20 min) 3) Interview (Time Frame: 45 min) 4)Modified Baecke Questionnaire (Time Frame: 30 min)
  For validation, the scores between the modified Baecke Questionnaire and the International Physical Activity Questionnaire (IPAQ) were compared and the correlation between Modified Baecke Questionnaire and VO2max (via Astrand-Rhyming Cycle Ergometer Test) and between modified Baecke Questionnaire and interview (via METS) were assessed.
  Tools:
  1. International Physical Activity
  2. Astrand-Rhyming Cycle Ergometer Test Questionnaires (VO2max)
  3. Interview (METS)
  2)

IPD SHARING:
Plan to Share IPD: No
GDPR protected

REFERENCES:
- [Derived] Stefanouli V, Kapreli E, Anastasiadi E, Nakastsis A, Strimpakos N. Validity and reliability of the Greek version of modified Baecke questionnaire. Public Health. 2022 Feb;203:58-64. doi: 10.1016/j.puhe.2021.11.017. Epub 2022 Jan 13. PMID 35032916